CLINICAL TRIAL: NCT03178292
Title: Conventional Antibiotic Prophylaxis Versus Add-On 5 Days Levofloxacin Before Percutaneous Nephrolithotomy (PCNL)
Brief Title: Conventional Antibiotic Prophylaxis Versus Add-On 5 Days Levofloxacin Before Percutaneous Nephrolithotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ab-PCNL
Record Dates: First submitted 2017-05-28; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Percutaneous Nephrolithotomy; Infection; Sepsis; Antibiotics
MeSH Terms: conditions — Infections; Sepsis | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levofloxacin (Active Comparator): Levofloxacin 500 mg daily for 5 days
  Interventions: Drug: Levofloxacin
- Placebo (Placebo Comparator): Placebo tab daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin 500Mg daily for 5 days
  Other Names: Levofloxacin 500Mg
  Arms: Levofloxacin
Drug: Placebo — Placebo Oral Tablet daily for 5 days
  Other Names: placebo Oral Tablet
  Arms: Placebo

SUMMARY:
To evaluate whether 5 days of levofloxacin before percutaneous nephrolithotomy (PCNL) in reducing upper urinary tract infection and urosepsis after PCNL.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is a minimally invasive procedure for removal of large volume upper urinary tract stones. Although PCNL is effective and yielding high stone-free rates, complications rates range from 18.30% to 83% with sepsis has been reported in 0.3% to 7.6% of cases result in the most common cause of perioperative mortality in PCNL patients.

Urosepsis after PNL is an important and potentially catastrophic complication. The overall incidence of fever (25%), bacteremia (23%), endotoxemia (34%) and septicemic shock occurs in 0.3%-2.5% of patients. Urosepsis and shock result from the intravasation of bacteria or endotoxins into bloodstream, which in turn increases with prolonged surgery, degree of hydronephrosis, bacterial load in the renal pelvis, and presence of infected stones.

Charton et al., concluded that without antibiotic prophylaxis 35% of patient suffered urinary tract infection a post-PCNL, although preoperative urine showing no growth. In a prospective but nonrandomized assessment of PCNL patients receiving oral ciprofloxacin, intravenous ciprofloxacin, or no antimicrobial treatment found postoperative urinary tract infection to occur in 17%, 0%, and 40% of patients, respectively. Mariappan et al., stated that midstream urine (MSU) culture does not represent upper tract infection in patients with obstructing stones. Also, stone and pelvic urine cultures are better predictors of upper tract infection and urosepsis in such cases.

Antibiotic prophylaxis has been recommended (Level of evidence: IIb, III) for patients subjected to PCNL to avert these infectious complications, as profiled in an American Urological Association (AUA) Best Practice Policy Statement. They also recommend antibiotic prophylaxis before shock wave lithotripsy and ureteroscopy with high level (Level of evidence: Ia and Ib, respectively) due to presence of meta-analysis and large randomised controlled trial.

The optimal timing, dosing, and duration of a prophylactic antibiotic regimen for PCNL procedures has also been a point of discussion. The AUA best practice policy statement currently recommends that a one-time dose on the day of the procedure is sufficient. The EAU guidelines are less definitive in concluding that a short course is adequate but that the "length of time is to be determined." Mariappan and colleagues in a prospective non-randomised trial found that 52 patients who had dilated collecting systems, stone burden greater than 2 cm, and no confounding factors predisposing to UTIs who received a 1-week course of ciprofloxacin before PCNL had a 3-fold lower risk of postoperative UTI and SIRS than 46 patients who received standard perioperative antibiotics on the day of surgery.

Bag and colleagues prospectively randomized 101 patients with greater than 2.5-cm kidney stones and/or hydronephrosis with sterile preoperative urine cultures to a 7-day course of nitrofurantoin versus no antibiotics before PCNL and found a statistically significant lower rate of postoperative SIRS (19% vs 49%), endotoxemia (18% vs 42%), positive result on kidney urine culture (0% vs 10%), and positive result on stone culture (8% vs 30%) in the arm receiving nitrofurantoin.

Although these two small series support a week of preoperative antibiotics before PCNL, larger, prospective, randomized studies are needed to better elucidate the risks and benefits of empiric antibiotics

ELIGIBILITY:
Inclusion Criteria:

* Stones ≥ 2.5 cm and/or hydronephrosis
* Sterile mid urine stream

Exclusion Criteria:

* Patients with a stent, nephrostomy tube or indwelling catheter
* Uncontrolled Diabetes mellitus
* Renal failure
* Fever before surgery
* Concomitant bladder stone or tumour
* Patients with active UTI
* Contralateral renal/ureteric stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2017-06-15 (Estimated); Study Completion 2017-06-15 (Estimated)

PRIMARY OUTCOMES:
Upper urinary tract infection and systemic inflammatory response syndrome (SIRS) after PCNL by Criteria for SIRS established by the American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference | 1 year
  SIRS if patient has Two or more of the 4 SIRS criteria

SECONDARY OUTCOMES:
difference between culture and sensitivity of Preoperative urine (MSU) and intraoperative renal pelvic urine and extracted stone. | 1 year
  Preoperative urine (MSU),intraoperative renal pelvic urine and extracted stone culture and sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shoma, MD, Study Chair — Urology and Nephrology center; Nasr Eltabey, MD, Study Director — Urology and Nephrology center; Mahmoud Laimon, Msc, Principal Investigator — Urology and Nephrology center; Muhamad Abdullateef, Msc, Principal Investigator — Urology and Nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes meta-analyses by contact the Prof. Ahmed Shoma, MD, Phd (Study Chair)